CLINICAL TRIAL: NCT05657262
Title: The Effect of Z Technique Treatment on Comfort, Pain and Undesirable Symptoms in Allergy Patients Receiving Immunotherapy: A Randomized Controlled Study
Brief Title: Effect of Z Technıque on Pain, Comfort, Symptoms in Ummunotherapy Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Gönül GÖKÇAY, Asist. Prof., Kafkas University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 81829502.903/94
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Immunotherapy
Keywords: Immunotherapy; Z technique; comfort; pain
MeSH Terms: conditions — Pain | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Intervention Model Description: experimental group: application of immunotherapy via Z technique control group: immunotherapy administration with standard procedure
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were divided into groups using the "simple randomization method". Participants were not informed about which group they belonged to. Automated computer-based randomization resulted in the execution of the experiment with the timing scenario and the confidential assignment of participants to one of the 2 intervention arms. The researcher was blind to all conditions until the participants started the computer program and the intervention began. Participants were also unaware of whether the group they were assigned to was an experimental or control condition. Additionally, researchers who code and analyze data will be blind to randomization and interference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experiment group will be applied with the Z technique. While applying the medicine with the Z technique, the tissue will be lifted with the thumb and forefinger of the left hand and pulled to the right, and the medicine will be slowly applied after the injector needle enters the tissue. When the application is finished, first the injector will be withdrawn, then the tissue will be released and the tissues will be restored (Altun, 2018).
  Interventions: Other: Pre-post test; Behavioral: experimental group
- Control group (Other): In the control group, the vaccine will be administered slowly with the standard technique.
  Interventions: Other: Pre-post test

INTERVENTIONS:
Other: Pre-post test — Personal Information Form, Vas Scale, Undesirable Symptoms Form and General Comfort Scale Questions will be asked to immunotherapy patients with this research.
Behavioral: experimental group — The experiment group will be applied with the Z technique.
  Arms: experimental group

SUMMARY:
An allergy is an abnormal response of the immune system to a generally harmless antigen. Pollens in the air play an important role in the formation of respiratory allergies and can be a trigger for the development of allergies (Won, 2022). By providing relaxation by nurses and taking measures to ensure the continuity of relaxation; Maintaining the well-being of the individual, family or society is possible with the comfort theory (Kolcaba and Kolcaba, 1991; Kolcaba, 1994). Although subcutaneous immunotherapy is performed in the presence of specialist physicians and trained nurses, some local side effects may develop after injection. One of the local side effects is pain, swelling and redness at the injection site (Arslan and Caliskaner, 2022).

The aim of this study; The aim of this study is to determine the effect of the treatment with the Z technique on allergy patients receiving immunotherapy on comfort, pain and adverse symptoms using a randomized controlled experimental method.

The hypotheses of the study H0: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy has no effect on comfort levels, pain and adverse symptoms H1: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy Has an Effect on Comfort Levels H2: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy Has an Effect on Pain Levels H3: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy Has an Effect on Undesirable Symptoms

DETAILED DESCRIPTION:
An allergy is an abnormal response of the immune system to a generally harmless antigen. Pollens in the air play an important role in the formation of respiratory allergies and can be a trigger for the development of allergies (Won, 2022). By providing relaxation by nurses and taking measures to ensure the continuity of relaxation; Maintaining the well-being of the individual, family or society is possible with the comfort theory (Kolcaba and Kolcaba, 1991; Kolcaba, 1994). Although subcutaneous immunotherapy is performed in the presence of specialist physicians and trained nurses, some local side effects may develop after injection. One of the local side effects is pain, swelling and redness at the injection site (Arslan and Caliskaner, 2022).

The aim of this study; The aim of this study is to determine the effect of the treatment with the Z technique on allergy patients receiving immunotherapy on comfort, pain and adverse symptoms using a randomized controlled experimental method.

The hypotheses of the study H0: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy has no effect on comfort levels, pain and adverse symptoms H1: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy Has an Effect on Comfort Levels H2: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy Has an Effect on Pain Levels H3: Treatment with Z Technique for Allergy Patients Receiving Immunotherapy Has an Effect on Undesirable Symptoms The research is a pre-post-test two-group randomized controlled study in experimental design.

The research population consists of 104 patients who received allergy treatment in Kocaeli Derince Training and Research Hospital in the last year. In this study, "G. In the calculation made using the "Power-3.1.9.2" program and using a similar study at the sample level at 80% confidence level (yilmaz et al., 2016), a total of 60 individuals, 30 of which were experimental and 30 of which were control, was determined.

ELIGIBILITY:
Inclusion Criteria:

To be receiving immunotherapy treatment at Kocaeli Derince Training and Research Hospital, be between the ages of 18-65, Volunteering to participate in the research,

Exclusion Criteria:

Not wanting to participate in the research voluntarily The state of moving the individual to a different country for any reason The end of the immunotherapy treatment period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
1.VAS Scale: | three months
  It is a scale numbered from 1 to 10 to measure the severity of pain that may occur after immunotherapy. Individuals rank 10 points for pain they feel most intensely and 1 point for pain they feel least severe.
2.General Comfort Scale: | three months
  Comfort Theory was developed by Katharina Kolcaba in 1990. The sub-dimensions of the General Comfort Scale, which was validated and reliable in Turkish by Çıtlık Sarıtaş et al. in 2018, were defined as relief (9 items), relaxation (9 items), and overcoming problems (10 items). The lowest possible value, 1, indicates low comfort, and the highest value, 6, indicates high comfort.
3. Undesirable Symptoms Tracking Form: | three months
  It is a form we developed to evaluate swelling, redness and leakage of the drug after 1 hour and 1 day after immunotherapy. Undesirable Symptoms Follow-up Form will be prepared and applied to the individuals participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül GÖKÇAY, Asist. Prof., Principal Investigator — Kafkas University-Kafkas University Faculty of Health Sciences; Zeynep Genç AKGÜN, RN, Study Chair — Derince Training and Research Hospital; Ayşe ÇEVİRME, Prof. Dr., Study Chair — Sakarya University-Sakarya University Faculty of Health Sciences; Aylin Meşe TUNÇ, MsC, Study Chair — Sakarya University-Sakarya University Faculty of Health Sciences; Nida EFETÜRK, Lecturer, Study Chair — Istanbul Okan University, Istanbul Okan University Vocational School of Health Services; Özge ERTÜRK, PhD, Study Chair — Sakarya University-Sakarya University Faculty of Health Sciences; Seda GÖĞER, Phd, Study Chair — Sakarya University-Sakarya University Health Care Services; Elif Seda UĞURLU, RN, Study Chair — Sakarya University Training and Research Hospital; Hülya İncirkuş KÜÇÜK, RN, Study Chair — Yalova State Hospital
Locations (1):
- Gönül GÖKÇAY, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is completed, it will be shared with all researchers.

REFERENCES:
- [Background] Kolcaba KY, Kolcaba RJ. An analysis of the concept of comfort. J Adv Nurs. 1991 Nov;16(11):1301-10. doi: 10.1111/j.1365-2648.1991.tb01558.x. PMID 1753026
- [Background] Kolcaba KY. A theory of holistic comfort for nursing. J Adv Nurs. 1994 Jun;19(6):1178-84. doi: 10.1111/j.1365-2648.1994.tb01202.x. PMID 7930099
- [Background] Yilmaz D, Khorshid L, Dedeoglu Y. The Effect of the Z-Track Technique on Pain and Drug Leakage in Intramuscular Injections. Clin Nurse Spec. 2016 Nov/Dec;30(6):E7-E12. doi: 10.1097/NUR.0000000000000245. PMID 27753676
- [Background] Arslan, Ş. & Çalışkaner, A. (2022) Subkutan Alerjen İmmünoterapisine Bağlı Lokal ve Sistemik Reaksiyonlar: Tek Merkezde 5 Yıllık Tecrübemiz. Kahramanmaraş Sütçü İmam Üniversitesi Tıp Fakültesi Dergisi, 17 (1) , 1-8 . DOI: 10.17517/ksutfd.839958.
- [Result] Oh JW. Pollen Allergy in a Changing Planetary Environment. Allergy Asthma Immunol Res. 2022 Mar;14(2):168-181. doi: 10.4168/aair.2022.14.2.168. PMID 35255535